CLINICAL TRIAL: NCT06620328
Title: Safety and Efficacy of Mechanical Versus Electrocautery Dilator for EUS-guided Biliary Drainage: A Prospective Randomized Controlled Trial
Brief Title: Safety and Efficacy of Mechanical Versus Electrocautery Dilator for EUS-guided Biliary Drainage (MED-BD)
Acronym: MED-BD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other); Taichung Veterans General Hospital (Other); Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other); Far Eastern Memorial Hospital (Other); China Medical University Hospital (Other); Chung Shan Medical University (Other); Taitung Mackay Memorial Hospital (Unknown); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other); Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202405138RINB
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-07

CONDITIONS: Biliary Obstruction
Keywords: Endoscopic ultrasound; Biliary drainage; Mechanical dilator; Electrocautery dilator; Interventional EUS

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Mechanical dilator (Experimental): Dilation of the needle tract is initially performed with an ultra-tapered mechanical dilator (7Fr ES Dilator; Zeon Medical Co., Tokyo, Japan).
  Interventions: Procedure: endoscopic ultrasonography-guided biliary drainage
- Electrocautery dilator (Active Comparator): Dilation of the needle tract is initially performed with a diathermic sheath (6Fr Cyst-Gastro set; Endoflex, Voerde, Germany).
  Interventions: Procedure: endoscopic ultrasonography-guided biliary drainage

INTERVENTIONS:
Procedure: endoscopic ultrasonography-guided biliary drainage — Skilled endosonographers performed EUS-BD with patients under conscious sedation by intravenous medication. All patients were given intravenous antibiotics prophylactically. A therapeutic curved linear array echoendoscope is positioned in the stomach with carbon dioxide insufflation. Standard 19G fine needles are used to puncture the dilated left intrahepatic bile duct or commo bile duct. Bile juice aspiration with 20ml syringe was performed to confirm intraductal puncture. After contrast medium injection, an insulated guidewire (0.025 inch VisiGlide2; Olympus Medical Systems, Tokyo, Japan) is advanced antegradely.
  Dilation of the needle tract is initially performed with a diathermic sheath (6Fr Cyst-Gastro set; Endoflex, Voerde, Germany) or an ultra-tapered mechanical dilator (7Fr ES Dilator; Zeon Medical Co., Tokyo, Japan) according to randomization result. If needed, additional dilation can be attempted with dilating balloon. Finally, the dedicated plastic stent or partially cover
  Other Names: EUS-BD

SUMMARY:
The purpose of this study is to investigate the likelihood of post-dilation bleeding using mechanical or electrocautery dilation. We hypothesized that the risk of bleeding is lower in the mechanical group.

DETAILED DESCRIPTION:
1. Study background In recent years, with the advancement of endoscopy, endoscopic ultrasound-guided biliary drainage (EUS-BD) has been increasingly applied in cases of failed endoscopic retrograde cholangiopancreatography(ERCP). According to the European Society of Gastrointestinal Endoscopy guidelines1, in patients with malignant obstruction of the distal bile duct, if ERCP drainage fails, EUS-guided biliary drainage is superior to percutaneous transhepatic biliary drainage (PTBD). In patients with malignant obstruction of the proximal bile duct combined with left-sided bile duct dilatation, EUS-guided biliary drainage can also be considered.

   The direct transmural technique is the most common method for EUS-guided biliary drainage.2,3 Under endoscopic ultrasound guidance, the dilated bile duct is observed from the stomach or duodenum. A fine needle is then used for duct puncture, and a guidewire is advanced into the duct followed by tract dilation to create an artificial fistula. Finally, a plastic or metal stent is placed to achieve drainage. Common complications of EUS-guided drainage procedures include bleeding, intestinal perforation, bile leakage, and stent migration, with tract dilation being the most common step leading to complications.4,5 The two main methods of tract dilation are electrocautery dilation and mechanical dilation. Currently, there are only retrospective studies comparing the success rates, complications, and short- and long-term outcomes between these two methods.6 However, no any randomized controlled trial has investigated the safety and efficacy of the two traction dilation method on EUS-BD. Therefore, this study will attempt to clarify the differences in bleeding, other complications, success rates of dilation, and drainage success rates between these two dilation methods through randomized allocation.
2. Study Design Multi-center randomized clinical trial (included National Taiwan University Hospital Hsin-Chu branch, National Cheng Kung University Hospital, Chang Gung Memorial Hospital, Taichung Veterans General Hospital, Taipei Tzu Chi Hospital, Shin Kong Wu Ho Su Memorial Hospital, Far Eastern Memorial Hospital, China Medical University Hospital, Chung Shan Medical University Hospital, and Taitung Mackay Memorial Hospital) will enroll 64 patients and the study period is 12 months.

   Randomization will be done by opening sealed opaque envelopes containing computer generated random sequences in blocks of 4.

   Patients will be randomly assigned to electrocautery dilation arm vs mechanical dilation arm on 1:1 basis.
3. Subjects Consecutive patients aged more than 18 years old indicated for EUS-guided biliary drainage were included.

   Inclusion criteria ： (1) Failed ERCP (2) The papilla is inaccessible owing to a surgically altered anatomy or gastric outlet obstruction (3) Contraindications for PTCD such as ascites and possibility of self-tube removal Exclusion criteria ： (1) Patients younger than 18 years old (2) Cancer infiltration of the gastric/duodenal wall within the planned puncture route (3) Patients with uncorrectable coagulopathy (4) Patients with unmanageable ascites (5) Patients with serious comorbidities that prohibited endoscopic management (6) Patients with pregnancy (7) Patients who cannot or refuse to provide informed consent
4. Study intervention Skilled endosonographers performed EUS-BD with patients under conscious sedation by intravenous medication. All patients were given intravenous antibiotics prophylactically. A therapeutic curved linear array echoendoscope is positioned in the stomach with carbon dioxide insufflation. Standard 19G fine needles are used to puncture the dilated left intrahepatic bile duct or commo bile duct. Bile juice aspiration with 20ml syringe was performed to confirm intraductal puncture. After contrast medium injection, an insulated guidewire (0.025 inch VisiGlide2; Olympus Medical Systems, Tokyo, Japan) is advanced antegradely.

   Dilation of the needle tract is initially performed with a diathermic sheath (6Fr Cyst-Gastro set; Endoflex, Voerde, Germany) or an ultra-tapered mechanical dilator (7Fr ES Dilator; Zeon Medical Co., Tokyo, Japan) according to randomization result. If needed, additional dilation can be attempted with dilating balloon. Finally, the dedicated plastic stent or partially covered self-expandable metallic stents (PCSEMS) is transmurally placed.
5. Measure outcomes

Primary outcome:

- Bleeding: hematemesis and/or melena or hemoglobin drop over 2g/dL, needed blood transfusion, endoscopic hemostasis, radiological intervention or surgery

Secondary outcomes:

* Tract dilation success: tract dilation was regarded as successful when the. maximum diameter portion of the first dilator into the bile duct.
* Final procedure success: a successful deployment of a stent in the intended location
* Procedural duration: the time elapsed between puncture of the intrahepatic duct and completion of deployment of stent
* Clinical success: a decrease in bilirubin within 30 days to < 75 % of levels before EUS-BD
* Recurrent biliary obstruction (RBO): cholangitis and jaundice accompanied by biliary dilation on imaging examinations
* Time to RBO (TRBO): the time from EUS-BD to the date of RBO occurrence
* Adverse events other than bleeding: pancreatitis, cholangitis, peritonitis, and perforation, in accordance with the American Society for GI Endoscopy lexicon7
* Length of hospital stay after procedure
* Overall survival

ELIGIBILITY:
Inclusion Criteria:

* Failed ERCP
* The papilla is inaccessible owing to a surgically altered anatomy or gastric outlet obstruction
* Contraindications for PTCD such as ascites and possibility of self-tube removal

Exclusion Criteria:

* Patients younger than 18 years old
* Cancer infiltration of the gastric/duodenal wall within the planned puncture route
* Patients with uncorrectable coagulopathy
* Patients with unmanageable ascites
* Patients with serious comorbidities that prohibited endoscopic management
* Patients with pregnancy
* Patients who cannot or refuse to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding | From randomization to four weeks after the procedure
  hematemesis and/or melena or hemoglobin drop over 2g/dL, needed blood transfusion, endoscopic hemostasis, radiological intervention or surgery

SECONDARY OUTCOMES:
Tract dilation success | From randomization to successful tract dilation using the first device (success), to using other dilation devices (fail) or to procedure termination (fail)
  tract dilation was regarded as successful when the maximum diameter portion of the first dilator into the bile duct.
Final procedure success | at the end of the procedure
  a successful deployment of a stent in the intended location
Procedural duration | between puncture of the intrahepatic duct and completion of deployment of stent
  the time elapsed between puncture of the intrahepatic duct and completion of deployment of stent
Clinical success | From enrollment to 30 days after procedure
  a decrease in bilirubin within 30 days to < 75 % of levels before EUS-BD
Time to Recurrent biliary obstruction | From the day of technically successful biliary drainage to the day of recurrent obstruction or to study completion an average of 1 year, whichever comes first
  the time from EUS-BD to the date of RBO occurrence
Overall survival | From date of randomization until the date of death from any cause or study completion, whichever came first, assessed up to 12 months
  The length of time from randomization to study completion that patients are still alive.
Length of hospital stay after procedure | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 12 months
  The number of days patients stay in the hospital
Adverse events other than bleeding | From the day of randomization to the date of death or through study completion, an average of 1 year
  pancreatitis, cholangitis, peritonitis, and perforation, in accordance with the American Society for GI Endoscopy lexicon

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Po Wang, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No